| <b>Document Type:</b> Statistical Analysis Plan | |
|---|---|
| Official Title: | A non-blinded retrospective biomarker add-on study to FIGARO-DKD for Bioprofiling the pharMacodynamic response to finerenone in FIGARO-DKD subjects (FIGARO-BM) |
| NCT Number: | NCT05013008 |
| <b>Document Date:</b> | 13 JUL 2022 |



#### BAY 94-8862 / 21952

# Title page

# A non-blinded biomarker add-on study to FIGARO-DKD for Bioprofiling the pharMacodynamic response to finerenone in FIGARO-DKD subjects (FIGARO-BM)

**Bayer study drug** BAY 94-8862 / Finerenone

**Study purpose:** Biomarker study

Clinical study III Date: 13 JUL 2022

phase:

**Study No.:** 21952 **Version:** 2.0

Author: PPD

#### **Confidential**

The information provided in this document is strictly confidential and is intended solely for the guidance of the clinical investigation. Reproduction or disclosure of this document, whether in part or in full, to parties not associated with the clinical investigation or its use for any other purpose without the prior written consent of the sponsor is not permitted.

Throughout this document, symbols indicating proprietary names (®, TM) are not displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.

This Statistical Analysis Plan is produced on a word-processing system and bears no signatures.

The approval of the Statistical Analysis Plan is documented in a separate Signature Document.

Reference Number: RD-SOP-1119 Supplement Version: 10

# Protocol No.: **BAY 94-8862 / 21952**

# **Table of Contents**

| Titl | e page | 1 |
|---|---|---|
| Tab | le of Tables | 2 |
| Abl | previations | 3 |
| 1. | Introduction | |
| 2. | Study Objectives | |
| 3. | Study Design | 4 |
| 4. | General Statistical Considerations | 4 |
| 4.1 | General Principles | 4 |
| 4.2 | Handling of Missing Data | |
| 4.3 | Interim Analyses and Data Monitoring | |
| 4.4 | Data Rules | 4 |
| <b>5.</b> | Analysis Sets | 5 |
| 6. | Statistical Methodology | 5 |
| 6.1 | Population characteristics | |
| 6.1. | • | |
| 6.1. | • | |
| 6.1. | | |
| 6.1. | 4 Prior and Concomitant Medication | 5 |
| 6.1. | Treatment duration, extent of exposure and compliance | 5 |
| 6.2 | Efficacy | 5 |
| 6.2. | 1 Main efficacy analysis | 6 |
| 6.3 | Pharmacokinetics/pharmacodynamics | 6 |
| 6.4 | Safety | 6 |
| 7. | Changes to the analyses specified in the study protocol | 6 |
| 8. | Document history and changes in the planned statistical analysis | 6 |
| 9. | References | |
| | Appendix | |
| 10.1 | 1 | |
| 10.2 | List of Biomarkers | 9 |
| Tab | le of Tables | |
| Tab | le 10-1 Estimated power for the primary endpoint | 8 |

Protocol No.: **BAY 94-8862 / 21952** 

#### **Abbreviations**

BFAS Biomarker Full Analysis Set gsd Geometric standard deviation

LOD Limit of Detection

mBFAS Modified Biomarker Full Analysis Set NPX Normalized Protein expression

QC Quality Check

SAP Statistical Analysis Plan sd Standard deviation

#### 1. Introduction

This statistical analysis plan describes a biomarker add-on study to the Phase 3 trial FIGARO-DKD (#17530). While the original trial, FIGARO-DKD, investigated the efficacy and safety of finerenone (a next-generation, non-steroidal mineralocorticoid-receptor antagonist [MRA]) on the reduction of cardiovascular morbidity and mortality in subjects with type 2 diabetes mellitus and the clinical diagnosis of diabetic kidney disease in addition to standard of care, this study (#21952) will solely perform exploratory biomarker analyses. All analyses will be done on existing leftover samples from selected FIGARO-DKD patients. Biomarkers described in this protocol (analytes) will be analyzed by novel proteomics technology (OLINK Explore®) allowing quantitative measurements of a multitude of markers in a small sample volume.

This SAP considers the main analysis of only 27 biomarkers as listed in section 10.2. Further analyses will be specified under separate cover in a biomarker analysis plan.

# 2. Study Objectives

Objectives and endpoints are listed in the table below:

| Objectives | Estimands/Endpoints |
|---|---|
| Primary | |
| To investigate long-term effect of<br>finerenone treatment, in addition to<br>standard-of-care, on circulating blood<br>biomarkers associated with fibrosis,<br>congestion, inflammation and vascular<br>function | Change in plasma biomarker levels after 36 months (Visit 11) of treatment versus 4 months (Visit 3) of treatment in a set of 27 pre-defined biomarkers (see section 10.2) |
| Other pre-specified | |
| To characterize mid- to long-term PD effects of finerenone and profiling the response to finerenone (vs placebo) in patients with DKD to describe biological pathways | Change in plasma biomarker levels after 12 months (Visit 5), 24 months (Visit 8) and 36 months (Visit 11), 48 months (Visit 14) 1 of treatment versus 4 months (Visit 3) of treatment |

Reference Number: RD-SOP-1119

<sup>&</sup>lt;sup>1</sup> Depending on availability of samples for visit

Protocol No.: **BAY 94-8862 / 21952** 

| • | To further investigate the study intervention and similar drugs (e.g. mode-of-action-related effects, safety) and to further investigate pathomechanisms deemed relevant to renal and cardiovascular diseases and associated health problems | • | Change in various biomarkers (e.g. diagnostic, safety, pharmacodynamic, monitoring, prognostic or potentially predictive biomarkers) |
|---|---|---|---|
| • | To assess relationship between | • | Change in biomarker levels at 12 months |
| | pharmacokinetics of finerenone and PD | | (Visit 5), 24 months (Visit 8) and 36 months |
| | effects | | (Visit 11) of treatment compared to exposure |

## 3. Study Design

Data from subjects consented under FIGARO-DKD (addendum approach) will be analyzed together with biomarker data acquired under FIGARO-BM.

The pooled data is intended to include approximately 600 (or more) FIGARO-DKD patients from 60 (or more) sites.

#### 4. General Statistical Considerations

## 4.1 General Principles

The statistical evaluation will be performed by using the software package SAS release 9.4 or higher (SAS Institute Inc., Cary, NC, USA). The main efficacy analysis will be performed in R on a validated server.

# 4.2 Handling of Missing Data

Missing data will not be imputed, unless otherwise specified.

#### 4.3 Interim Analyses and Data Monitoring

Not applicable.

#### 4.4 Data Rules

The QC-flag, which is provided by OLINK, will be coded in a four-digit-code according to the table below:

| | Value = 0 | Value = 1 | Description |
|---|---|---|---|
| 1 <sup>st</sup> digit | Data point passed OLINKs QC-metrics | Data point failed some of OLINKs QC-metrics | Pass/Fail of OLINKs predefined QC metrics |
| 2 <sup>nd</sup> digit | No outlier | Outlier | Outlier status, based on PCA |
| 3 <sup>rd</sup> digit | No outlier | Outlier | Outlier status, based on NPX median and range |
| 4 <sup>th</sup> digit | NPX > LOD | NPX < LOD | Above limit of detection or not |

Data, which is QC-flagged by OLINKs predefined QC metrics (i.e. value = 1 in the first digit), will be set to missing for all analyses.

Visit 3 data will be considered as baseline measurements.

Demographic and baseline characteristics will be obtained from the FIGARO-DKD data.

NPX data is on log<sub>2</sub>-scale.

For further data rules, refer to the FIGARO-DKD SAP.

Reference Number: RD-SOP-1119

Protocol No.: **BAY 94-8862 / 21952** 

## 5. Analysis Sets

#### BFAS (Biomarker Full Analysis Set):

All participants with valid informed consent for this biomarker study and which meet study enrollment criteria as defined in the study protocol.

#### mBFAS (modified Biomarker Full Analysis Set):

All participants with valid informed consent for this biomarker study, which meet the following criteria:

- Study enrollment criteria as defined in the study protocol.
- Analyzed biomarker samples at Visit 3 (4 months) and Visit 11 (36 months). Biomarker samples that were shipped at ambient temperatures were not analyzed.
- On Treatment at Visit 3 (4 months) and Visit 11 (36 months).

# 6. Statistical Methodology

## 6.1 Population characteristics

Population characteristics from FIGARO-DKD will be repeated for the modified Biomarker Full Analysis Set. Detailed information on the respective analyses are described in the FIGARO-DKD SAP.

#### 6.1.1 Disposition

The number of subjects overall as well as by treatment group, region, country and study site will be repeated for the mBFAS.

#### 6.1.2 Demography and baseline characteristics

The demographic and other baseline characteristics tables will be repeated for the mBFAS. For these tables the baseline definition of FIGARO-DKD will be used instead of Visit 3.

## 6.1.3 Medical history

The medical history tables will be repeated for the mBFAS.

#### 6.1.4 Prior and Concomitant Medication

The prior and concomitant medication tables will be repeated for the mBFAS.

#### 6.1.5 Treatment duration, extent of exposure and compliance

The treatment duration, extent of exposure and compliance tables will be repeated for the mBFAS.

#### 6.2 Efficacy

All efficacy analyses will be performed on the 27 biomarkers listed in section 10.2. The remaining biomarkers analysed in the OLINK panel will only be included as prior information for the moderated t-test.

Reference Number: RD-SOP-1119

Protocol No.: **BAY 94-8862 / 21952** 

## 6.2.1 Main efficacy analysis

The primary efficacy variable is the change in plasma biomarker levels after 36 months (Visit 11) of treatment versus 4 months (Visit 3) of treatment of subjects on treatment at both visits. The NPX differences (corresponding to log-transformed ratio to baseline) of biomarker levels will be analysed for the set of 27 pre-defined biomarkers in treatment group compared to placebo, based on the modified Biomarker Full Analysis Set (mBFAS) as defined in section 5.

The hypotheses ' $H_0^i$ :  $\beta_i = 0$ ' (i=1,...,27) will be tested at a two-sided significance level of 5%, where  $\beta_i$  is the estimator for the difference in log-transformed ratios of biomarker levels of Visit 11 to Visit 3 between treatment and placebo group for the i-th of the 27 pre-specified biomarkers. The analysis will be adjusted for a selection of baseline characteristics and strafication factors. The selection of the adjustment covariates is related to the biomarker pre-processing of OLINK. The p-values obtained from the moderated t-statistics [1] testing the difference between treatment and placebo group on the log-transformed ratios of biomarker levels from Visit 11 to Visit 3, based on the OLINK Explore 1536 panel, will be adjusted for multiple testing according to Benjamini and Hochberg [2]. According to this method the false discovery rate can be controlled by ordering the 27 p-values  $p_i$  (i=1,...,27) by ascending value and comparing the i-th p-value with the adjusted significance level of  $\frac{i}{27}$  · 5% respectively.

Alternatively the *i*-th p-value  $p_i$  can be adjusted as min  $\left(\left(\min_{j\geq i}\frac{27}{j}\cdot p_i\right),1\right)$ , as described by Benjamini, Heller and Yekutieli [3].

The study will be considered as successful if at least one adjusted p-value is below the significance level of 5%.

Summary statistics and line plots (geometric mean with geometric standard deviation [gsd]-error bars over time) as well as boxplots for the ratio of Visit 11 to Visit 3 will be generated.

# 6.3 Pharmacokinetics/pharmacodynamics

Not applicable.

#### 6.4 Safety

Not applicable.

# 7. Changes to the analyses specified in the study protocol

According to the protocol, the primary endpoint should be analyzed in the Biomarker Full Analysis Set (BFAS) including all subjects with signed informed consent. As the analysis is only feasible, if also a biomarker is measured, an new analysis set was defined including subjects with signed informed consent and a biomarker measurement. The primary analysis will be conducted in this modified Biomarker Full Analysis Set (mBFAS).

# 8. Document history and changes in the planned statistical analysis

SAP version 0.1 dated 08 DEC 2021 submitted for internal review

SAP version 0.2 dated 11 FEB 2022 submitted for internal review

Approved SAP version 1.0 dated 06 APR 2022

Reference Number: RD-SOP-1119

Protocol No.: **BAY 94-8862 / 21952** 

#### Approved SAP supplement version 2.0 dated 13 JUL 2022

- As delivery of second batch of biomarkers will take place earlier than expected, all biomarkers will be included in the primary analysis as described in the protocol, instead of only the first batch as described in SAP version 1.0.
- Added coding-table of OLINKs QC-flag, which was not available for SAP v. 1.0.
- Added statement on scale of NPX data.
- Added more detailed description of Benjamini-Hochberg procedure.

#### 9. References

- [1] G. Smyth, "Linear models and empirical Bayes methods for assessing differential expression in microarray experiments," in *Statistical Application in Genetics and Molecular Biology. vol 3*, Melbourne, 2004, pp. 1-26.
- [2] H. Y. Benajmini Y, "Controlling the false discovery rate: a practical and powerful approach to multiple testing.," *Journal of the Royal Statistical Society Series B*, *57*, pp. 289-300, 1995.
- [3] Y. Benjamini, R. Heller and D. Yekutieli, "Selective inference in complex research," *Philosophical Transactions of the Royal Society*, vol. 367, pp. 1-17, 2009.

Reference Number: RD-SOP-1119 Supplement Version: 10 Protocol No.: **BAY 94-8862 / 21952** 

# 10. Appendix

## **10.1** Determination of sample size

Table 10-1 summarizes the results of a power simulation based on the following assumptions:

- Two sided test, significance level of 5%.
- Beneficial effect of finerenone on 4 of the 27 biomarkers with a ratio of biomarker levels from Visit 11 to Visit 3 (month 4) under finerenone of 10%, 15% or 20% compared to placebo.
- Inter-subject variability of 25% (geometric standard deviation of 1.25)
- Intra-subject variability from Visit 3 to Visit 11 of 20% (geometric standard deviation of 1.2)
- Assay-variability of 10% (geometric standard deviation of 1.1)

Table 10-1 Estimated power for the primary endpoint

| Treatment effect size | Number of subjects per arm | Power to detect<br>4 biomarkers | Power to<br>detect 3<br>biomarkers<br>or more | Power to<br>detect 2<br>biomarkers<br>or more | Power to detect<br>1 biomarkers or more |
|---|---|---|---|---|---|
| 10% | 75 | 2.5% | 5.4% | 9.5% | 16.8% |
| | 100 | 4.5% | 9.2% | 15.2% | 24.2% |
| | 250 | 26.4% | 42.0% | 55.2% | 67.4% |
| | 300 | 37.4% | 55.4% | 66.9% | 77.4% |
| | 400 | 57.6% | 74.4% | 83.6% | 90.3% |
| 15% | 75 | 13.4% | 24.3% | 34.9% | 48.0% |
| | 100 | 24.2% | 39.3% | 51.8% | 63.8% |
| | 250 | 86.1% | 94.8% | 97.7% | 99.2% |
| | 300 | 94.2% | 98.8% | 99.5% | 99.9% |
| | 400 | 99.4% | 100.0% | 100.0% | 100.0% |
| 20% | 75 | 45.0% | 62.4% | 74.0% | 83.4% |
| | 100 | 67.3% | 82.0% | 89.5% | 94.3% |
| | 250 | 99.9% | 100.0% | 100.0% | 100.0% |
| | 300 | 100.0% | 100.0% | 100.0% | 100.0% |
| | 400 | 100.0% | 100.0% | 100.0% | 100.0% |

Power estimations are based on the methodology described in section 9.4 and Monte-Carlo simulations with 10,000 iterations per scenario.Numbers in bold indicate the anticipated number of subjects per arm (total subjects = 600). Greyshading indicates a power of ≥80%

As shown in Table 10-1, the intended patient number of 600 with 300 subjects per arm (finerenone and placebo 1:1) would lead to a power of 94.2% to correctly detect all 4 biomarkers with beneficial effect at an estimated effect size of 15% between visit 3 (4 months) and visit 11 (36 months). For description of the panels refer to the study protocol. All simulations concerning sample size determination were conducted using R.

Reference Number: RD-SOP-1119

Protocol No.: **BAY 94-8862 / 21952** 

# 10.2 List of Biomarkers

| Uniprot | Protein name | Gene name |
|---------|------------------------------------------------------|-----------|
| P07911 | Uromodulin | UMOD |
| Q03167 | Transforming growth factor beta receptor type 3 | TGFBR3 |
| O15467 | C-C motif chemokine 16 | CCL16 |
| P02452 | Collagen alpha-1 | COL1A1 |
| P04275 | von Willebrand factor | VWF |
| P05121 | Plasminogen activator inhibitor 1 // PAI-1 | SERPINE1 |
| P16581 | E-selectin | SELE |
| Q9H2A7 | C-X-C motif chemokine 16 | CXCL16 |
| Q9UBP4 | Dickkopf-related protein 3 | DKK3 |
| P01033 | Metalloproteinase inhibitor 1 | TIMP1 |
| Q16627 | C-C motif chemokine 14 | CCL14 |
| P15144 | Aminopeptidase N | ANPEP |
| Q99969 | Retinoic acid receptor responder protein 2 | RARRES2 |
| P07585 | Decorin | DCN |
| P09237 | Matrilysin // MMP7 | MMP7 |
| Q03405 | Urokinase plasminogen activator surface receptor | PLAUR |
| P29279 | CCN family member 2 // CTGF | CCN2 |
| Q13219 | Pappalysin-1 | PAPPA |
| P01137 | Transforming growth factor beta-1 proprotein | TGFB1 |
| Q13261 | Interleukin-15 receptor subunit alpha | IL15RA |
| P35442 | Thrombospondin-2 | THBS2 |
| P14780 | Matrix metalloproteinase-9 | MMP9 |
| P19438 | Tumor necrosis factor receptor superfamily member 1A | TNFRSF1A |
| P13500 | C-C motif chemokine 2 // / MCP-1 | CCL2 |
| P12931 | Proto-oncogene tyrosine-protein kinase Src | SRC |
| P02760 | Protein AMBP | AMBP |
| O95388 | WNT1-inducible-signaling pathway protein 1 //CCN4 | WISP1 |

Reference Number: RD-SOP-1119 Supplement Version: 10